CLINICAL TRIAL: NCT02150928
Title: An Open-Label, Single-Arm, Multicenter Pharmacokinetic Study of Intramuscular Erwinaze® (Asparaginase Erwinia Chrysanthemi)/Erwinase® (Crisantaspase) Administered Following Hypersensitivity to E. Coli Asparaginase in Young Adults With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Brief Title: An Open-Label, Single-Arm, Multicenter Pharmacokinetic Study of Intramuscular Erwinaze® (Asparaginase Erwinia Chrysanthemi)/Erwinase® (Crisantaspase)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-006
Record Dates: First submitted 2014-05-21; First posted 2014-05-30 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)/Lymphoblastic Lymphoma (LBL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant

ARMS (1):
- Erwinaze / Erwinase (Experimental)
  Interventions: Drug: Erwinaze® (Asparaginase Erwinia Chrysanthemi)/Erwinase® (Crisantaspase)

INTERVENTIONS:
Drug: Erwinaze® (Asparaginase Erwinia Chrysanthemi)/Erwinase® (Crisantaspase) — * Enrolled patients will receive asparaginase Erwinia chrysanthemi 25,000 IU/m2 administered intramuscularly (IM) on a Monday/Wednesday/Friday schedule (all dosing regimens will start on a Monday)
  * All patients will receive at least 1 course (2 weeks) of treatment with asparaginase Erwinia chrysanthemi (1 course=6 doses), and a maximum number of courses needed to complete their remaining asparaginase therapy (up to 15 courses)
  * Eligible patients may not begin treatment with asparaginase Erwinia chrysanthemi until their serum asparaginase activity level is below the assay detectable limit

SUMMARY:
The purpose of this study is to evaluate the serum asparaginase activity in subjects ages 18 to <40 years with ALL or LBL who have developed a hypersensitivity to native E. coli asparaginase or pegaspargase.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of ALL or LBL
2. Be 18 to <40 years of age at the time of enrollment
3. Have a documented ≥ Grade 2 clinical hypersensitivity reaction to native E. coli asparaginase (e.g., Elspar or Kidrolase) or pegaspargase (Oncaspar)
4. Have the following asparaginase doses remaining in their treatment plan:

   * At least two (2) consecutive weeks of native E. coli asparaginase treatment OR
   * At least one (1) dose of pegaspargase (Oncaspar)
5. Have a direct bilirubin ≤ Grade 2 (<3.0 mg/dL [52 µmol/L])
6. Have amylase and lipase within normal limits (per institutional standards)
7. Have a serum asparaginase activity below the detectable limit during screening prior to the first dose of study drug (Erwinaze)
8. Consent to use a medically acceptable method of contraception throughout the entire study period and for 4 weeks after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or the partner include abstinence, birth control pills or patches, diaphragm and spermicide, condom and vaginal spermicide, surgical sterilization, postmenopausal, vasectomy (>6 months prior to baseline), and progestin implant or injection.
9. Have signed informed consent

Exclusion Criteria:

1. Prior history of ≥ Grade 3 pancreatitis
2. Prior history of a major thrombotic event as assessed by the investigator, or any subject with a history of asparaginase-associated serious hemorrhagic or thrombotic event requiring prolonged anticoagulation therapy with agents such as heparin
3. Prior treatment with Erwinaze
4. Pregnant or lactating female subjects or female subjects of childbearing potential not willing to use an adequate method of birth control (listed above) for the duration of the study
5. Subjects with a history of human immunodeficiency virus (HIV) or hepatitis.
6. Any other condition that would cause a risk (in the investigator's judgment) to subjects if they participate in the trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Serum asparaginase activity levels | 48 h postdose 5

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Bergstrom, Md, PhD, Study Director — Jazz Pharamceuticals
Locations (1):
- Hospital of Navarra, Pamplona, Navarre, Spain